CLINICAL TRIAL: NCT06977425
Title: Efficacy of Intraoperative Magnesium Sulphate vs Dexmedetomidine on Emergence Agitation in Pediatric Patients Under Sevoflurane Anesthesia
Brief Title: Efficacy of Intraoperative Magnesium Sulphate vs Dexmedetomidine on Emergence Agitation in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Esraa medhat Ezzat Mohamed, Resident of Anesthesia, Intensive Care and Pain Management, Faculty of Medicine, Ain Shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU MS112/2024
Record Dates: First submitted 2025-04-04; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Magnesium Sulphate; Dexmedetomidine; Emergence Agitation; Pediatric Patients
MeSH Terms: conditions — Emergence Delirium | interventions — Magnesium Sulfate; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium sulphate group (Experimental): Patients received an initial intravenous loading dose of 30 mg/kg of 10% magnesium sulfate solution over 10 min. This will be followed by a continuous infusion of (10mg/kg/hr) for the entire duration of surgery.
  Interventions: Drug: Magnesium sulphate
- Dexmedetomidine group (Experimental): Patients received dexmedetomidine infusion 0.5 μg/kg over 10 min as a bolus dose, followed by 0.2 μg/kg/h all over the operation.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Magnesium sulphate — Patients received an initial intravenous loading dose of 30 mg/kg of 10% magnesium sulfate solution over 10 min. This will be followed by a continuous infusion of (10mg/kg/hr) for the entire duration of surgery.
  Arms: Magnesium sulphate group
Drug: Dexmedetomidine — Patients received dexmedetomidine infusion 0.5 μg/kg over 10 min as a bolus dose, followed by 0.2 μg/kg/h all over the operation.
  Arms: Dexmedetomidine group

SUMMARY:
This study aimed to compare the effectiveness of intraoperative magnesium sulfate versus dexmedetomidine infusions on emergence agitation that follows anesthesia using sevoflurane immediately and after 30 min in the post-anesthesia care unit (PACU), regarding Pediatric Anesthesia Emergence Delirium Scale (PAED), Richmond agitation sedation scale (RASS), and hemodynamics

DETAILED DESCRIPTION:
Emergence agitation (EA) is a postoperative phenomenon that occurs in children after sevoflurane anesthesia, with an occurrence rate of up to 80%.

Dexmedetomidine acts on α-2 adrenergic receptors, producing sedation and hypnosis with anxiolytic effects, without a clinically significant depressive impact on heart rate, blood pressure, and respiratory rate, complementing an earlier study suggesting the possible effective and safe use of dexmedetomidine as a part of anesthesia care to prevent emergence agitation in children.

Magnesium sulfate also has been reported to decrease the incidence and severity of Emergence agitation and the need for postoperative rescue doses of analgesia in children, and its use was not associated with increased postoperative side effects or delayed recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age from 4 to 8 years old.
* Both sexes.
* Patients American Society of Anesthesiologists (ASA) Physical Status I to II.
* Duration of surgery: not exceeding two hours

Exclusion Criteria:

* Legal guardian refusal.
* Neurological abnormalities, such as cerebral palsy.
* Any physical and/or developmental challenge.
* Patients on sedatives, anticonvulsants, or any medications that may alter conscious level in children.
* Coexisting renal or cardiovascular diseases.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Pediatric Anesthesia Emergence Delirium Scale | 30 minutes postoperatively
  Pediatric Anesthesia Emergence Delirium Scale (PAED). The PAED Scale consists of five characteristics that are each scored by using a 5-point Likert scale:
  * The child makes eye contact with the caregiver
  * The child is aware of his or her surroundings
  * The child's actions are purposeful,
  * The child is restless
  * The child is inconsolable We set the threshold score for the presence of pediatric emergence delirium using the PAED Scale at a score higher than or equal to 10 based on the sensitivity and specificity reported in the literature.

SECONDARY OUTCOMES:
Richmond agitation sedation scale (RASS) | 30 minutes postoperatively
  The Richmond agitation sedation scale (RASS) assesses five levels of sedation:
  * (5) unarousable with no response to voice or physical stimulation
  * (4) deep sedation with no response to voice but movement to physical stimuli
  * (3) moderate sedation with movement to voice but no eye contact
  * (2) light sedation and briefly awakens (ie, less than 10 seconds) with eye contact to voice
  * (1) drowsy (ie, not fully alert) but has sustained (ie, more than 10 seconds) awakening with eye contact to voice
Heart rate | 30 minutes postoperatively
  Heart rate will be recorded from the start of injection till 30 minutes postoperatively.
Blood pressure | 30 minutes postoperatively
  Blood pressure will be recorded from the start of injection till 30 minutes postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.